CLINICAL TRIAL: NCT03653728
Title: Non-invasive Neuro-monitoring for Head Injury: Use of Near Infra-red Spectroscopy for Early Detection of Delayed Intracranial Haematoma
Brief Title: Near Infra-red Spectroscopy for Detection of Intracranial Haematoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. David Yuen Chung CHAN, Neurosurgery Resident, Chinese University of Hong Kong
Other Study IDs: NTEC-2018-0106
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Traumatic Brain Injury; Intracerebral Hemorrhage
Keywords: non-invasive monitoring; near-infrared spectroscopy; traumatic brain injury; cerebral contusion
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Hemorrhage; Brain Contusion | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Traumatic brain injury with cerebral contusions
  Interventions: Device: Near infrared spectroscopy

INTERVENTIONS:
Device: Near infrared spectroscopy — All patients would be receiving the same treatment including application of non-invasive monitoring with near-infrared spectroscopy (NIRS) together with the standard of care with interval CT Brain scan for all patients.
  Non-invasive monitoring with near-infrared spectroscopy (NIRS) is very safe and is in current daily routine clinical use for intraoperative patients.

SUMMARY:
Fall with head injury is becoming an epidemic challenge especially with the ageing population. Contributing factors for mortality and poor functional outcome included development of cerebral contusion and delayed traumatic intracerebral haematoma. There is a higher prevalence especially with the increasing use of antiplatelets and anticoagulants.

Non-invasive monitoring such as near-infrared spectroscopy (NIRS) is sensitive in detecting intracranial changes. The role and efficacy of this non-invasive method has not been specifically established in patients with head injury as an initial non-operative monitoring. This is particular important in the setting of a general ward in which nursing staff is limited. The advantages of these noninvasive monitoring might have a role of continuous neuro-monitoring. They can also potentially reduce the number of unnecessary repeated CT Brain in the context of limited radiology staff and resources. Timely detection and treatment of this condition accordingly is crucial. Potential options of non-invasive monitoring such as nearinfrared spectroscopy (NIRS) is to be investigated.

The aim of this study is to determine the sensitivity and specificity of NIRS as a non-invasive monitoring in detecting delayed intracranial injuries in comparison with the Gold Standard CT Brain. Study design is Prospective sensitivity and specificity study of Near Infra-red Spectroscopy (NIRS) as a non-invasive monitoring in detecting delayed intracranial injuries in comparison with the Gold Standard CT Brain in Hong Kong Chinese. Consecutive patients admitted to Prince of Wales Hospital, Hong Kong would be recruited. Outcome measures including correlation of non-invasive monitoring with near-infrared spectroscopy (NIRS) to CT Brain findings including any increase in haematoma size, cerebral edema or mass effect. Secondary outcome including 30 days mortality and functional outcome at 3 months.

DETAILED DESCRIPTION:
Introduction: Fall with head injury is becoming an epidemic challenge especially with the ageing population. Contributing factors for mortality and poor functional outcome included development of cerebral contusion and delayed traumatic intracerebral haematoma. There is a higher prevalence especially with the increasing use of antiplatelets and anticoagulants.

Non-invasive monitoring such as near-infrared spectroscopy (NIRS) is sensitive in detecting intracranial changes. The role and efficacy of this non-invasive method has not been specifically established in patients with head injury as an initial non-operative monitoring. This is particular important in the setting of a general ward in which nursing staff is limited. The advantages of these non-invasive monitoring might have a role of continuous neuro-monitoring. They can also potentially reduce the number of unnecessary repeated CT Brain in the context of limited radiology staff and resources.

Timely detection and treatment of this condition accordingly is crucial. Potential options of non-invasive monitoring such as near-infrared spectroscopy (NIRS) is to be investigated.

Aims and Hypotheses to be tested:

The aim of this study is to determine the sensitivity and specificity of near-infrared spectroscopy (NIRS) as a non-invasive monitoring in detecting delayed intracranial injuries in comparison with the Gold Standard CT Brain.

Plan of Investigation:

This is a prospective sensitivity and specificity correlation study of Near Infra-red Spectroscopy (NIRS) as a non-invasive monitoring in detecting delayed intracranial injuries in comparison with the Gold Standard CT Brain in Hong Kong Chinese. Consecutive patients admitted to Prince of Wales Hospital, Hong Kong would be recruited.

Consecutive patients fulfilling the inclusion and exclusion criteria are treated with standard of care with near-infrared spectroscopy (NIRS). Criteria to proceed for repeat CT Brain scan 1) clinical deterioration of GCS >2 points, 2) NIRS monitoring has increase in difference in absorbance of light at 760nm >0.3, or 3) 8 hours after admission for baseline interval scan for all patients as part of the standard of care. Non-invasive monitoring with near-infrared spectroscopy (NIRS) would be applied to all patients' forehead for consecutively 48 hours after admission.

Inclusion criteria

1. Age greater than or equal to 18 years old,
2. History of traumatic brain injury,
3. Radiological evidence of intracranial haematoma,
4. Glasgow Coma Scale (GCS) less than 15 upon admission,
5. Not undergoing immediate operation,
6. Admission to the general ward or high dependence unit of Neurosurgery, Prince of Wales Hospital.

Exclusion criteria

1. Presence of frontal scalp laceration preventing the application of non-invasive monitoring on the forehead,
2. Presence of pneumocephale,
3. Requirement of immediate surgical intervention as judged by the on-call neurosurgeon.
4. Patients who have joined other drug trial in the last four weeks;
5. Pregnant or on breast feeding;
6. Any other reasons that the researchers consider unsuitable.

Primary outcome - Correlation coefficient of near-infrared spectroscopy (NIRS) to CT Brain findings including any increase in haematoma size, cerebral edema or mass effect.

Secondary outcomes

- Secondary outcome including number of CT scan performed, correlation of NIRS reading with Glasgow coma scale (GCS), rate of intervention with either medical treatment such as use of mannitol, Transamin or blood product transfusion, or surgical treatment such as operation, 30 days mortality and functional outcome at 3 months.

Purpose and Potential:

Near-infrared spectroscopy (NIRS) can offer continuous neuro-monitoring. This is particular important in the setting of a general ward in which nursing staff is limited. This allows early detection of delayed haematoma for early intervention. At the same time, the use of NIRS can potentially reduce the number of unnecessary repeated CT Brain in the context of limited radiology staff and resources.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years old,
2. History of traumatic brain injury,
3. Radiological evidence of intracranial haematoma,
4. Glasgow Coma Scale (GCS) less than 15 upon admission,
5. Not undergoing immediate operation,
6. Admission to the general ward or high dependence unit of Neurosurgery, Prince of Wales Hospital.

Exclusion Criteria:

1. Presence of frontal scalp laceration preventing the application of non-invasive monitoring on the forehead,
2. Presence of pneumocephale,
3. Requirement of immediate surgical intervention as judged by the on-call neurosurgeon.
4. Patients who have joined other drug trial in the last four weeks;
5. Pregnant or on breast feeding;
6. Any other reasons that the researchers consider unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive traumatic brain injury patients fulfilling the inclusion and exclusion criteria are treated with standard of care with near-infrared spectroscopy (NIRS).
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient | 1 week
  Correlation coefficient of near-infrared spectroscopy (NIRS) to CT Brain findings including any increase in haematoma size, cerebral edema or mass effect.

SECONDARY OUTCOMES:
30 days mortality | 30 days
  30 days mortality
modified Rankin Scale | 3 months
  modified Rankin Scale (mRS) at 3 months. The mRS scale ranges from 0 to 6, in which 0 indicates no disability, while 6 indicates death.

OTHER OUTCOMES:
correlation of NIRS reading with Glasgow coma scale (GCS) | 1 week
  correlation of NIRS reading with Glasgow coma scale (GCS). The scale GCS ranges from 3 to 15, in which a GCS of 3 indicates a status of deep coma, whereas a GCS of 15 indicates a fully conscious status.
Number of CT performed | 1 week
  Number of CT performed
Other intervention such as blood product transfusion or operation | 1 week
  Other intervention such as blood product transfusion or operation

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Neurosurgery, Department of Surgery, Prince of Wales Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folkerson LE, Sloan D, Cotton BA, Holcomb JB, Tomasek JS, Wade CE. Predicting progressive hemorrhagic injury from isolated traumatic brain injury and coagulation. Surgery. 2015 Sep;158(3):655-61. doi: 10.1016/j.surg.2015.02.029. Epub 2015 Jun 9. PMID 26067457
- [Background] Oertel M, Kelly DF, McArthur D, Boscardin WJ, Glenn TC, Lee JH, Gravori T, Obukhov D, McBride DQ, Martin NA. Progressive hemorrhage after head trauma: predictors and consequences of the evolving injury. J Neurosurg. 2002 Jan;96(1):109-16. doi: 10.3171/jns.2002.96.1.0109. PMID 11794591
- [Background] Narayan RK, Maas AI, Servadei F, Skolnick BE, Tillinger MN, Marshall LF; Traumatic Intracerebral Hemorrhage Study Group. Progression of traumatic intracerebral hemorrhage: a prospective observational study. J Neurotrauma. 2008 Jun;25(6):629-39. doi: 10.1089/neu.2007.0385. PMID 18491950
- [Background] Alahmadi H, Vachhrajani S, Cusimano MD. The natural history of brain contusion: an analysis of radiological and clinical progression. J Neurosurg. 2010 May;112(5):1139-45. doi: 10.3171/2009.5.JNS081369. PMID 19575576
- [Background] Weigl W, Milej D, Janusek D, Wojtkiewicz S, Sawosz P, Kacprzak M, Gerega A, Maniewski R, Liebert A. Application of optical methods in the monitoring of traumatic brain injury: A review. J Cereb Blood Flow Metab. 2016 Nov;36(11):1825-1843. doi: 10.1177/0271678X16667953. Epub 2016 Sep 7. PMID 27604312
- [Background] Kim B, Jeong H, Kim J, Kim T, Kim K, Lee H, Ahn S, Jo YH, Lee JH, Hwang JE. Incidence and risk factors of delayed intracranial hemorrhage in the emergency department. Am J Emerg Med. 2018 Feb;36(2):271-276. doi: 10.1016/j.ajem.2017.08.009. Epub 2017 Aug 4. PMID 28811212
- [Background] Chieregato A, Fainardi E, Morselli-Labate AM, Antonelli V, Compagnone C, Targa L, Kraus J, Servadei F. Factors associated with neurological outcome and lesion progression in traumatic subarachnoid hemorrhage patients. Neurosurgery. 2005 Apr;56(4):671-80; discussion 671-80. doi: 10.1227/01.neu.0000156200.76331.7a. PMID 15792505
- [Background] Chang EF, Meeker M, Holland MC. Acute traumatic intraparenchymal hemorrhage: risk factors for progression in the early post-injury period. Neurosurgery. 2006 Apr;58(4):647-56; discussion 647-56. doi: 10.1227/01.NEU.0000197101.68538.E6. PMID 16575328
- [Background] Poon WS, Wong GK, Ng SC. The quantitative time-resolved near infrared spectroscopy (TR-NIRs) for bedside cerebrohemodynamic monitoring after aneurysmal subarachnoid hemorrhage: can we predict delayed neurological deficits? World Neurosurg. 2010 May;73(5):465-6. doi: 10.1016/j.wneu.2010.03.029. No abstract available. PMID 20920925
- [Background] Gomersall CD, Leung PL, Gin T, Joynt GM, Young RJ, Poon WS, Oh TE. A comparison of the Hamamatsu NIRO 500 and the INVOS 3100 near-infrared spectrophotometers. Anaesth Intensive Care. 1998 Oct;26(5):548-57. doi: 10.1177/0310057X9802600512. PMID 9807611
- [Background] Gomersall CD, Joynt GM, Gin T, Freebairn RC, Stewart IE. Failure of the INVOS 3100 cerebral oximeter to detect complete absence of cerebral blood flow. Crit Care Med. 1997 Jul;25(7):1252-4. doi: 10.1097/00003246-199707000-00031. No abstract available. PMID 9233756